CLINICAL TRIAL: NCT00006221
Title: A Phase I Study of BMS-247550 (NSC 710428) Given Weekly X 3 Every 4 Weeks in Patients With Advanced Malignancies
Brief Title: BMS-247550 in Treating Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068141; UTHSC-IDD-99-32; SACI-IDD-99-32; NCI-150
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2004-07

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ixabepilone

ARMS (1):
- Arm I (Experimental): Patients receive BMS-247550 IV over 1 hour once weekly on weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of BMS-247550 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at that dose level. Patients treated at the MTD receive treatment once weekly on weeks 1-3 of each 4-week course.
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
Phase I trial to study the effectiveness of BMS-247550 in treating patients who have malignant solid tumors or lymphoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of BMS-247550 in patients with advanced malignancies.

II. Determine the qualitative and quantitative toxic effects of this regimen in these patients.

III. Determine the pharmacokinetics and pharmacodynamics of this regimen in these patients.

IV. Determine the antitumor effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to prior therapy (heavily pretreated vs minimally pretreated).

Patients receive BMS-247550 IV over 1 hour once weekly on weeks 1-4. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BMS-247550 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at that dose level. Patients treated at the MTD receive treatment once weekly on weeks 1-3 of each 4-week course.

Patients are followed within 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor or lymphoma for which no other potentially curative therapeutic option exists or demonstrates increased survival (considering tumor type, stage, and number of prior regimens)
* No symptomatic brain metastases requiring dexamethasone

  * No progression or cerebral edema on CT scan or MRI within the past 4 weeks

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Hemoglobin at least 8.5 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No atrial or ventricular arrhythmias requiring medication
* No ischemic event within the past 6 months

Other:

* No pre-existing peripheral neuropathy greater than grade 1
* No other serious medical illness or active infection that would preclude study participation
* No dementia, psychiatric illness, or other alteration in mental status that would preclude study compliance
* No other active malignancy except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No history of allergy or hypersensitivity reaction to paclitaxel or other Cremophor EL-containing compound
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study completion

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since prior anticancer hormonal therapy and recovered
* No concurrent hormonal therapy except LHRH agonists for non-castrated prostate cancer, contraceptives, hormone replacement therapy (e.g., conjugated estrogens), or megestrol as an appetite stimulant

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* Concurrent palliative radiotherapy to limited sites allowed

Surgery:

* At least 4 weeks since prior surgery and recovered

Other:

* At least 30 days since prior investigational agents and recovered
* No other concurrent experimental medications
* No concurrent antiretroviral (HAART) therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2000-11; Primary Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris H. Takimoto, MD, PhD, FACP, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (3):
- United States (3):
  - Cancer Therapy and Research Center, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas